CLINICAL TRIAL: NCT04169165
Title: How to Improve Patient Compliance for Metabolic Evaluation and Medical & Dietary Prophylaxis in Calcium Stone Patients?
Brief Title: Patient Compliance for Metabolic Evaluation and Medical Management in Calcium Stone Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: EULIS Colloborative Research Working Group (Network)
Responsible Party: Sponsor
Other Study IDs: eCORE-S-19-001
Record Dates: First submitted 2019-11-16; First posted 2019-11-19 (Actual); Last update posted 2019-11-19 (Actual); Status verified 2019-11

CONDITIONS: Kidney Calculi; Nephrolithiasis; Patient Compliance; Calcium Oxalate Urolithiasis
Keywords: kidney stone; calcium oxalate stone; patient compliance; nephrolithiasis
MeSH Terms: conditions — Kidney Calculi; Nephrolithiasis; Patient Compliance; Nephrolithiasis, Calcium Oxalate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- compliant patients: Patients with compliance to suggestions on metabolic evaluation and dietary/medical advices
- non-compliant patient: Patients without compliance to suggestions on metabolic evaluation and dietary/medical advices

SUMMARY:
Calcium oxalate stone, the most common type worldwide, has a recurrence rate of around 50% in ten years. Therefore, identifying the underlying pathophysiological aspects via metabolic evaluation and suggestions for medical & dietary prophylaxis in calcium stone patients is of upmost importance.

However, one of the greatest problem with metabolic evaluation and subsequent therapeutic advices is the patient compliance. Therefore, it is important to identify factors related to patient compliance for metabolic evaluation and medical & dietary prophylaxis in calcium stone patients

DETAILED DESCRIPTION:
Nephrolithiasis is an important health problem that can deteriorate the renal functions in long term and affects the patients' quality of life. One of the major problems about renal stones is the high rate of recurrence. Calcium oxalate stone, the most common type worldwide, has a recurrence rate of around 50% in ten years. Therefore, identifying the underlying pathophysiological aspects via metabolic evaluation and suggestions for medical & dietary prophylaxis in calcium stone patients is of upmost importance.

However, one of the greatest problem with metabolic evaluation and subsequent therapeutic advices is the patient compliance. In the previous studies, even in case of a dedicated stone clinic, the drop out rate for preventive measures were over 37% per year. The patients' non-compliance may be related to a number of factors associated with the stone clinic, demographic characteristics of the patients, past medical history of the patients, and even the recommended tests and the therapeutic advices.

Therefore, it is important to identify factors related to patient compliance for metabolic evaluation and medical & dietary prophylaxis in calcium stone patients

Methods:

Parameters to be recorded

Age Gender Level of education

* of stone episodes
* of surgical intervention Type of surgical intervention History of SWL Concomitant diseases Other medications Type of metabolic evaluation (24 hour urine, spot morning urine, serum etc.) Drug for medical prophylaxis Dosage of medication (bid/tid, etc.) Side effects Dietary recommendations Compliance to metabolic evaluation Compliance to medical treatment

Statistics:

Patients will be grouped based on:

compliance to metabolic evaluation compliance to medical treatment

The parameters listed above will be compared between the groups with univariate analysis (logistic regression).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of calcium oxalate kidney stones
* Suggested metabolic evaluation for kidney stone
* Suggested dietary and/or medical treatment for kidney stone
* Accepted participation in the study

Exclusion Criteria:

* Age less than 18
* Mental disorders

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients diagnosed with a calcium oxalate kidney stones and suggested for metabolic evaluation and dietary and/or medical management will be enrolled in the study.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2020-01 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2021-02 (Estimated)

PRIMARY OUTCOMES:
patient compliance rate of metabolic evaluation | 30 days
  the rate of the patients undergo metabolic evaluation tests will be determined
patient compliance rate of dietary suggestions | 6 months
  the rate of the patients that follow the dietary suggestions will be determined
patient compliance rate of drug treatments | 6 months
  the rate of the patients that have the prescribed drugs will be determined

SECONDARY OUTCOMES:
factors associated with non-compliance to metabolic evaluation | 3 months
  the factors that are related to poor patient compliance to metabolic evaluation will be determined in multivariate analysis
factors associated with non-compliance to dietary suggestions | 3 months
  the factors that are related to poor patient compliance to dietary suggestions will be determined in multivariate analysis
factors associated with non-compliance to medications | 3 months
  the factors that are related to poor patient compliance to medications will be determined in multivariate analysis

IPD SHARING:
Plan to Share IPD: No
All centers will enter their data for every single patient to an online database. The participating centers will be provided a username and a password to enter to the system. All centers will see the data of their own patients and only the number of patients enrolled from other centers.

REFERENCES:
- [Result] Hess B. Renal stone clinic survey: calcium stone formers' self-declared understanding of and adherence to physician's recommendations. Urolithiasis. 2017 Aug;45(4):363-370. doi: 10.1007/s00240-016-0916-3. Epub 2016 Aug 29. PMID 27573100
- [Result] Prezioso D, Strazzullo P, Lotti T, Bianchi G, Borghi L, Caione P, Carini M, Caudarella R, Ferraro M, Gambaro G, Gelosa M, Guttilla A, Illiano E, Martino M, Meschi T, Messa P, Miano R, Napodano G, Nouvenne A, Rendina D, Rocco F, Rosa M, Sanseverino R, Salerno A, Spatafora S, Tasca A, Ticinesi A, Travaglini F, Trinchieri A, Vespasiani G, Zattoni F; CLU Working Group. Dietary treatment of urinary risk factors for renal stone formation. A review of CLU Working Group. Arch Ital Urol Androl. 2015 Jul 7;87(2):105-20. doi: 10.4081/aiua.2015.2.105. PMID 26150027
- [Result] Trinchieri A. Diet and renal stone formation. Minerva Med. 2013 Feb;104(1):41-54. PMID 23392537
- [Result] Skolarikos A, Straub M, Knoll T, Sarica K, Seitz C, Petrik A, Turk C. Metabolic evaluation and recurrence prevention for urinary stone patients: EAU guidelines. Eur Urol. 2015 Apr;67(4):750-63. doi: 10.1016/j.eururo.2014.10.029. Epub 2014 Nov 20. PMID 25454613
- [Result] Bensalah K, Tuncel A, Raman JD, Bagrodia A, Pearle M, Lotan Y. How physician and patient perceptions differ regarding medical management of stone disease. J Urol. 2009 Sep;182(3):998-1004. doi: 10.1016/j.juro.2009.05.025. Epub 2009 Jul 18. PMID 19616801
- [Result] Parks JH, Asplin JR, Coe FL. Patient adherence to long-term medical treatment of kidney stones. J Urol. 2001 Dec;166(6):2057-60. PMID 11696706
- [Result] Dauw CA, Yi Y, Bierlein MJ, Yan P, Alruwaily AF, Ghani KR, Wolf JS Jr, Hollenbeck BK, Hollingsworth JM. Medication Nonadherence and Effectiveness of Preventive Pharmacological Therapy for Kidney Stones. J Urol. 2016 Mar;195(3):648-52. doi: 10.1016/j.juro.2015.10.082. Epub 2015 Oct 17. PMID 26485048
- [Result] Pietrow P, Auge BK, Weizer AZ, Delvecchio FC, Silverstein AD, Mathias B, Albala DM, Preminger GM. Durability of the medical management of cystinuria. J Urol. 2003 Jan;169(1):68-70. doi: 10.1016/S0022-5347(05)64037-2. PMID 12478105